CLINICAL TRIAL: NCT04940052
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Dabrafenib Plus Trametinib in Previously Treated Patients With Locally Advanced or Metastatic, Radio-active Iodine Refractory BRAFV600E Mutation-positive Differentiated Thyroid Cancer (DTC)
Brief Title: Study of Efficacy and Safety of Dabrafenib in Combination With Trametinib in Previously Treated Patients With Metastatic, Radio-active Iodine Refractory BRAF V600E Mutation Positive Differentiated Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDRB436J12301
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Differentiated Thyroid Cancer (DTC)
Keywords: Differentiated Thyroid Cancer (DTC); Locally advanced or metastatic differentiated thyroid cancer; radio active iodine refractory; previously targeted therapy; B-Raf proto-oncogene, serine/threonine kinase (BRAF); BRAFV600E mutation; Dabrafenib (DRB436); trametinib (TMT212)
MeSH Terms: interventions — dabrafenib; trametinib

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 2:1 ratio to either dabrafenib plus trametinib or placebo. Patients will be stratified by number of prior VEGFR targeted therapy (1 versus 2) and prior Lenvatinib treatment (yes versus no).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dabrafenib plus Trametinib (Experimental): Eligible participants will receive Dabrafenib 150 mg twice a day (BID) and Trametinib 2 mg once a day (QD) until disease progression as per RECIST 1.1 as confirmed by blinded independent review committee (BIRC), unacceptable toxicity, pregnancy, loss of clinical benefit as determined by the investigator, withdrawal of consent, lost to follow-up, death, or study termination by the sponsor.
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Dabrafenib Placebo plus Trametinib Placebo (Placebo Comparator): Eligible participants will receive matching placebo for Dabrafenib 150 mg twice a day (BID) and matching placebo for Trametinib 2 mg once a day (QD) until disease progression as per RECIST 1.1 as confirmed by blinded independent review committee (BIRC), unacceptable toxicity, pregnancy, loss of clinical benefit as determined by the investigator, withdrawal of consent, lost to follow-up, death, or study termination by the sponsor.
  Interventions: Drug: Trametinib Placebo; Drug: Dabrafenib placebo

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib 150 mg capsule administered orally twice a day (BID)
  Other Names: DRB436
  Arms: Dabrafenib plus Trametinib
Drug: Trametinib — Trametinib 2 mg tablet administered once a day (QD)
  Other Names: TMT212
  Arms: Dabrafenib plus Trametinib
Drug: Trametinib Placebo — matching placebo tablet for Trametinib 2 mg will be administered orally once a day (QD)
  Arms: Dabrafenib Placebo plus Trametinib Placebo
Drug: Dabrafenib placebo — matching placebo capsule for Dabrafenib 150 mg will be administered orally twice a day (BID)
  Arms: Dabrafenib Placebo plus Trametinib Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of dabrafenib in combination with trametinib for treating adult patients with locally advanced or metastatic Differentiated Thyroid Cancer (DTC) harboring the BRAFV600E mutation, who are refractory to radioactive iodine (RAI) therapy and have experienced disease progression following one or two prior VEGFR-targeted treatments.

DETAILED DESCRIPTION:
This is a global, multicenter, randomized, double-blind, placebo-controlled phase III study to evaluate the efficacy and safety of dabrafenib plus trametinib in adult patients with locally advanced or metastatic BRAFV600E mutation-positive, differentiated thyroid carcinoma who are refractory to radioactive iodine and have progressed following prior VEGFR targeted therapy. The scientific objective guiding the primary estimand is based on the Progression Free Survival (PFS) as per BIRC assessment using RECIST 1.1 criteria.

Patients randomized in the placebo arm for whom disease progression as per RECIST 1.1 is confirmed by Blinded Independent Review Committee (BIRC) and who meet the eligibility criteria outlined in the study protocol will be given the option to crossover to the open-label dabrafenib plus trametinib treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent
* Male or female ≥ 18 years of age at time of informed consent
* Histologically or cytologically confirmed diagnosis of advanced/metastatic differentiated thyroid carcinoma
* Radioactive-iodine refractory disease
* BRAF V600E mutation-positive tumor sample as per central laboratory result
* Has progressed on at least 1 but not more than 2 prior VEGFR targeted therapies
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* At least one measurable lesion as defined by RECIST v1.1.

Key Exclusion Criteria:

* Anaplastic or medullary carcinoma of the thyroid
* Previous treatment with a BRAF inhibitor and/or a MEK inhibitor
* Concomitant RET Fusion-Positive Thyroid Cancer
* Treatment with any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before randomization
* Treatment with any type of anticancer antibody (including investigational antibody) or systemic chemotherapy within 4 weeks before randomization
* Treatment with radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before randomization
* A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy

Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2027-06-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From randomization to first documented progression or deaths, whichever comes first, assessed up to approximately 2 years
  Progression Free Survival (PFS) was defined as the time from the date of randomization to the date of the first documented progression according to RECIST 1.1 based on Blinded Independent Review Committee (BIRC) assessment, or death due to any cause.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From randomization up to approximately 2 years
  Overall Response Rate (ORR) was defined as the proportion of participants with Best Overall Response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), as per Blinded Independent Review Committee (BIRC) assessment and according to RECIST 1.1.
Overall Survival (OS) | From randomization to death assessed up to approximately 5 years
  Overall Survival (OS) is defined as the time from the date of randomization to the date of death due to any cause.
Duration of Response (DOR) | From the start date of the first documented response of complete response or partial response and the date defined as the date of the first documented progression or death due to any cause up to 2 years
  Duration of Response (DOR) applied only to patients whose Best Overall Response (BOR) was a confirmed Complete Response (CR) or Partial Response (PR), as determined by the Blinded Independent Review Committee (BIRC) assessment according to RECIST 1.1. The start date was defined as the date of the first documented confirmed CR or PR, and the end date corresponded to the date of the first documented confirmed progression or death from any cause. Patients who remained without progression or death from any cause were censored at the date of their last adequate tumor assessment prior to the initiation of any new antineoplastic therapy.
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Throughout study completion, an average 5 years
  The distribution of adverse events will be conducted through the analysis of frequencies for treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs), based on the monitoring of relevant clinical and laboratory safety parameters. Treatment-emergent adverse events (TEAEs) in this study will be defined as events that begin after the first dose of study treatment and continue until 30 days after the last dose, or events that are present prior to the first dose and increase in severity based on preferred term within 30 days following the last dose.
Number of participants with trametinib associated serous retinopathy ocular events | screening, week 4, week 8, week 12, week 20 and every 12 weeks after week 20, up to approximately 2 years
  Standard ophthalmic examinations were performed by an ophthalmologist, and Optical Coherence Tomography (OCT) was conducted at mandated visits. Analysis of the optical coherence tomography data was carried out to evaluate the incidence, type, and severity of trametinib-associated serous retinopathy ocular events.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (36):
- United States (2):
  - Northwestern University Med School, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Brazil (3):
  - Novartis Investigative Site, Rio de Janiero, Rio de Janeiro
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, London, Ontario
- China (13):
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Xuzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- India (3):
  - Novartis Investigative Site, Hisar, Haryana
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Chennai
- Malaysia (3):
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Edirne, Merkez
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Adana, Yuregir
- Novartis Investigative Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.